CLINICAL TRIAL: NCT00168181
Title: A Phase III Randomized Trial Comparing Oral Pilocarpine (Salagen) Versus Submandibular Salivary Gland Transfer Protocol, For the Prevention of Radiation (XRT) Induced Xerostomia in Head and Neck Cancer Patients
Brief Title: Trial Comparing Oral Pilocarpine (Salagen) Versus Submandibular Salivary Gland Transfer Protocol, For the Prevention of Radiation (XRT) Induced Xerostomia in Head and Neck Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alberta Health services (Other)
Collaborators: CancerCare Manitoba (Other); Jewish General Hospital (Other); Newfoundland Cancer Treatment & Research Foundation (Unknown); Notre-dame Hospital (Unknown); Ottawa Hospital Research Institute (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HN-04-0010
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Cancer; Head and Neck Cancer
Keywords: salagen; gland transfer; randomized; xerostomia
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms; Xerostomia | interventions — Pilocarpine

INTERVENTIONS:
Procedure: Submandibular gland Transfer
Drug: Salagen

SUMMARY:
This is a study to see whether the drug Salagen or salivary gland transfer is better for the prevention of dryness of the mouth in patients with head and neck cancer receiving radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated and confirmed histological diagnosis of squamous cell/adenoid cystic carcinoma of the oropharynx, hypopharynx, larynx, and patients with unknown primary tumor with metastases to the neck nodes and squamous cell carcinoma of the skin of head and neck region with ipsilateral neck nodes (more than one node) metastases.
2. Radiation volume to encompass > or equal to 80% of major salivary glands (parotids and the non-transferred submandibular salivary gland) and have > or equal to 50 Gys delivered to that volume via external beam.
3. Karnofsky performance score > or equal to 70
4. Minimum age 18 years
5. The patient must sign a study-specific informed consent prior to study entry
6. Expected survival > or equal to one year

Exclusion Criteria:

1. Carcinoma of nasopharynx, oral cavity, N3 disease, bilateral neck node involvement, pre-epiglottic space involvement, involvement of level 1 nodes on either side of the neck, and patients with post-operative recurrent disease.
2. Salivary gland malignancy
3. Salivary gland disease
4. Use of anti-cholinergic drugs and tricyclic drugs
5. Delay in XRT of more than 8 weeks following the curative surgery
6. Pregnant or lactating females are not eligible. Patients of childbearing potential should agree to use an effective method of contraception
7. Prior head and neck irradiation
8. Recurrent disease
9. Allergy to pilocarpine
10. Patients with uncontrolled asthma, acute iritis, or narrow angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2002-04; Study Completion 2008-04

PRIMARY OUTCOMES:
To compare the efficacy of prevention of XRT induced xerostomia using two different approaches: oral Pilocarpine versus submandibular salivary gland transfer protocol; To compare the rate and severity of XRT induced xerostomia using these two strategies

SECONDARY OUTCOMES:
To evaluate the incidence of oral candidiasis, percutaneous endoscopic gastrostomy (PEG), and hospitalization during XRT

CONTACTS AND LOCATIONS:
Overall Officials: Naresh Jha, MBBS, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada